CLINICAL TRIAL: NCT06377917
Title: The IMPACT Trial: Investigating Micro-Manipulation Procedures for Assisted Hatching Timing
Brief Title: Investigating Micro-Manipulation Procedures for Assisted Hatching Timing
Acronym: IMPACT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2304-BRG-057-JF
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cleavage Stage Assisted Hatching (AH) (Other): Current standard of care. Day 3 or cleavage stage embryos will have the zona pellucida hatched with a laser.
  Interventions: Other: Laser Assisted Hatching
- Blastocyst Stage Assisted Hatching (AH) (Experimental): Blastocyst stage embryos on day 5,6 or 7 will have the zona pellucida hatched with a laser.
  Interventions: Other: Laser Assisted Hatching

INTERVENTIONS:
Other: Laser Assisted Hatching — Routine assisted hatching procedure will be performed on both groups at the different embryo developmental phases.

SUMMARY:
This study aims to assess the clinical significance of cleavage stage (Day 3) assisted hatching compared to assisted hatching at the blastocyst stage (Day 5,6,7) of embryo development at the time of trophectoderm (TE) biopsy for patients undergoing in vitro fertilization (IVF) and preimplantation genetic testing for aneuploidy (PGT-A) for treatment of their infertility.

DETAILED DESCRIPTION:
The proposed study aims to perform a split cohort study where each patient's cohort of fertilized zygotes, (two pronuclei or 2PNs) is split into two groups and randomized, thus allowing each patient to serve as their own control and decreasing confounding variables. Half of the cohort will proceed with the current standard of day 3 or cleavage assisted hatching and the other half of the cohort will receive the sequential hatching and trophectoderm biopsy procedure at the blastocyst stage of embryo development.

ELIGIBILITY:
Inclusion Criteria for participants:

1. Patients undergoing an IVF cycle with plan for subsequent FET of a single euploid embryo
2. <4 2PNs prior to randomization
3. Female partners age <42 years old at start of VOR cycle
4. Normal ovarian reserve:

   1. AMH ≥ 1.2 ng/mL
   2. AFC ≥ 8
   3. FSH ≤ 12IU/L
5. BMI <38
6. Patients who desire to transfer the best quality embryo for their embryo transfer.

Exclusion Criteria for participants:

1. All patients who do not voluntarily give their written consent for participation
2. Patients with a prior failed IVF cycle - defined as no blastocysts
3. Patients with a history of more than one failed euploid embryo transfer
4. Donor oocyte cycles
5. Gestational Carriers
6. Male partner with <100,000 total motile spermatozoa per ejaculate (donor sperm is acceptable)
7. Use of surgical procedures to obtain sperm
8. Communicating hydrosalpinges without a plan for surgical correct prior to frozen embryo transfer
9. Endometrial Insufficiency, as defined by a prior cycle with maximal endometrial thickness <6mm,), or persistent endometrial fluid
10. Single gene disorders, chromosomal translocations, or any other disorders requiring a more detailed embryo genetic analysis than standard PGT-A

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Blastulation Rate | 1 week after vaginal oocyte retrieval (VOR)
  Blastulation rate per 2 pronuclei (PN) in each group

SECONDARY OUTCOMES:
Embryo morphologic grade | 1 week post VOR
  Gardner and Modified Gardner grading system will be used
Timing of blastulation | 1 week post VOR
  proportion of blastocysts that blastulate on day 5,6 or 7
Aneuploidy rate | 2 weeks post blastulation
  Rates of whole chromosome positive and negative preimplantation genetic testing (PGT-A) results
Positive pregnancy rate | approximately 9 days post embryo transfer
  proportion of positive pregnancy tests per embryo transfer
Sustained implantation rate | 8-9 weeks gestational age or approximately 5-6 weeks post embryo transfer
  proportion of patients discharged with presence of a fetal heartbeat
Pregnancy loss rate | approximately 1-2 months post initial bHCG
  proportion of pregnancy patients who experience a loss of pregnancy
Live birth rate | approximately 40 weeks gestation or 7 months post discharge
  proportion of patients who deliver a live born infant

CONTACTS AND LOCATIONS:
Overall Officials: Jason Fransiak, MD, Principal Investigator — Reproductive Medicine Associates of New Jersey
Locations (1):
- Reproductive Medicine Associates of New Jersey, Marlton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No